CLINICAL TRIAL: NCT03071848
Title: Retrospective Multicenter Observational Study to Evaluate Safety and Effectiveness of Bevacizumab (Avastin®) in Combination With Paclitaxel and Cisplatin/Carboplatin or Toptecan in Patients With Advanced Cervical Cancer
Brief Title: A Study to Evaluate Safety and Effectiveness of Bevacizumab in Combination With Paclitaxel and Cisplatin/Carboplatin or Toptecan in Participants With Advanced Cervical Cancer
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML39360
Record Dates: First submitted 2017-03-02; First posted 2017-03-07 (Actual); Last update posted 2018-03-16 (Actual); Status verified 2018-03

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Bevacizumab: Participants with advanced cervical cancer (metastatic, recurrent or persistent) who have received treatment with bevacizumab from 01 January 2015 to 01 January 2016 (retrospective and independent from this study) combined with standard chemotherapy (cisplatin/carboplatin or topotecan and paclitaxel) will be observed.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — This was an observational study.

SUMMARY:
This study will evaluate the safety of bevacizumab (Avastin®) combined with standard chemotherapy in participant with advanced cervical cancer, with special focus on the incidence of gastrointestinal (GI) and genitourinary (GU) fistulas and GI perforations in the common practice setting.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Diagnosis of primary stage IVB, recurrent or persistent squamous cell carcinoma, adenosquamous carcinoma, or adenocarcinoma of the cervix which is not amenable to curative treatment with surgery and/or radiation therapy
* Retrospective clinical decision made to initiate therapy with bevacizumab (Avastin®) combined with standard chemotherapy (cisplatin or carboplatin or topotecan and paclitaxel) between 01 January 2015 and 01 January 2016
* All participants must have received at least one dose of bevacizumab combined with standard chemotherapy between 01 January 2015 and 01 January 2016 AND have at least 12 months of documented follow up, from treatment start, unless died or lost to follow up within the minimum study entry follow up period
* Availability of documentation of for advanced cervical cancer (including prior treatment as applicable) and follow up in the participant's medical records

Exclusion Criteria:

* Participation during the study period in an interventional clinical trial or any other interventional study that may impact advanced cervical cancer outcome
* Participants who have received prior therapy with any anti-VEGF drug, including bevacizumab

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with advanced cervical cancer (metastatic, recurrent or persistent) who have received treatment with bevacizumab from 01 January 2015 to 01 January 2016 will be observed.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2017-04-06 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Gastrointestinal (GI) and Genitourinary (GU) Fistulas and GI Perforations | Up to 12 months
  Participants with GI and GU fistulas and GI perforation events will be reported according to Common Terminology Criteria for Adverse Events (CTCAE V4.0).

SECONDARY OUTCOMES:
Percentage of Participants who Received Radiotherapy Prior to GI and GU Fistulas and GI Perforation Events | Up to 12 months
  Participants who received radiotherapy prior to GI and GU fistulas and GI perforation events will be reported.
Percentage of Participants who Received Internal, External and Other Radiotherapy | Up to 12 months
  Participants who received internal, external and other radiotherapy will be reported. External radiotherapy will include "Non Precision Orientated" that includes classic cobalt or "Precision Orientated" that includes Linear accelerator.
Number of Doses of Prior Radiotherapy | Up to 12 months
  Doses of prior radiotherapy will be reported.
Percentage of Participants With Selected Adverse Events of Special Interest (AESIs) | Up to 12 months
  Adverse events of special interest (AESI) for this study included: hypertension, proteinuria, wound healing complication, bleeding /haemorrrhage (including pulmonary haemorrhage and CNS bleeding), arterial and venous thromboembolic events (ATES; VTES), congestive heart failure (CHF), posterior reversible encephalopathy syndrome (PRES), fistula/abscess (other than genitourinary and gastrointestinal), gastrointestinal perforations and gallbladder perforation.
Overall Response Rate (ORR) | Up to 12 months
  Overall response rate was defined as the percentage of participants who had confirmed complete response (CR) or partial response (PR). CR is defined as disappearance of all target and non-target lesions. PR is defined as at least a 30% decrease in the sum of longest dimensions (LD) of all target measurable lesions taking as reference the baseline sum of LD. There can be no unequivocal progression of non-target lesions and no new lesions. In the case where the only target lesion is a solitary pelvic mass measured by physical exam, which is not radiographically measurable, a 50% decrease in the LD is required.
Progression Free Survival (PFS) | Up to 12 months
  PFS is defined as the time from the first dose of treatment to the first occurrence of progression, or death from any cause as assessed by the investigator. Progressive disease (PD): at least a 20% increase in the sum of LD target lesions taking as reference the smallest sum LD recorded since study entry.
Overall Survival (OS) | Up to 12 months
  OS is defined as the time from the first dose of treatment to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (12):
- Argentina (12):
  - Hospital General de Agudos Juan Antonio Fernandez, Buenos Aires
  - Hospital General de Agudos J. A. Penna ; Breast Pathology, Buenos Aires
  - Instituto Ángel H. Roffo - Universidad de Buenos Aires, Buenos Aires
  - Hospital Julio C. Perrando, Chaco
  - Centro Oncologico Riojano Integral (CORI), La Rioja
  - Hospital Interzonal General De Agudos "Luisa C. de Gandulfo", Lomas de Zamora
  - Hospital Privado de Comunidad; Oncology, Mar del Plata
  - Hosp Provincial D. Centenarios; Oncology Dept, Rosario
  - CENICLAR, Rosario
  - Policlínico regional de San Luis, San Luis
  - Centro Medico San Roque, San Miguel de Tucumán
  - Hospital Pablo Soria, San Salvador de Jujuy